CLINICAL TRIAL: NCT03872856
Title: Home Blood Pressure Monitoring Intervention for Self-Management of High Blood Pressure Among Alaska Native People
Brief Title: Blood Pressure-Improving Control Among Alaska Native People" (BP-ICAN)
Acronym: CHAR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southcentral Foundation (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, Denise Dillard, Director of Research, Southcentral Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP-ICAN-1U54MD011240-01; 2017-08-038 (Other: Alaska Area Institutional Review Board)
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Alaska Native and American Indian; Home Blood Pressure Monitoring; Self-efficacy; Primary Care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Group randomized comparison trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BP-ICAN (Active Comparator): Participants in the BP-ICAN arm will receive a home blood pressure monitor to be used twice daily for 12 months. Participants' home blood pressure measurements will be shared with their provider and participants will receive a series of text messages including topics on the importance of managing hypertension, reminders to measure blood pressure with their device, and motivational messages on diet and exercise.
  Interventions: Device: BP-ICAN
- Control (No Intervention): Participants in the control arm will receive care as usual for the treatment of hypertension

INTERVENTIONS:
Device: BP-ICAN — One of two home blood pressure monitor devices will be used.
  1. Omron 7 Series Wrist cuff
  2. Omron 10 Series Upper Arm cuff
  Arms: BP-ICAN

SUMMARY:
"Blood Pressure: Improving Control among Alaska Native People" (BP-ICAN) that targets blood pressure control among Alaska Native and American Indian (AN/AI) people diagnosed with hypertension. Participants will include adults with a diagnosis of hypertension who have not achieved blood pressure control. Primary Care Center (PCC) provider teams and associated panels of Alaska Native or American Indian (ANAI) adults will be randomized into the control or intervention arm. The investigators will recruit up to 10 ANAI adults per PCC provider for a total of 324 participants. Intervention participants will receive a home blood pressure monitor (HBPM), upload personal home blood pressure values into a data mall, and be encouraged to communicate with providers and pharmacists about HBPM results using an online electronic health record application, telephone, or other existing clinical processes. HBPM measurements for each intervention arm participant will be provided to provider teams and integrated pharmacists. Control participants will receive care as usual. Data will be collected over a 12 month period. Participants will meet with investigators at time of consent (baseline), and 3, 6, and 12 months after baseline. At each visit, participants will have blood pressure measured using 3 methods (aneroid sphygmomanometer, automated Omron upper arm cuff device, and automated Omron wrist cuff device), complete surveys, and have height, weight, and arm circumference measured. In-person measures are omitted during the pandemic and only one method of blood pressure measurement is used (upper arm cuff device). Clinical and service utilization information will be electronically queried with participant consent. The investigators will examine whether participants in the intervention arm have better blood pressure control at the end of the 12 month period than participants in the control arm.

DETAILED DESCRIPTION:
Background:

Cardiovascular disease (CVD) and stroke have become leading causes of mortality among ANAI people, who experience CVD disparities in incidence, risk factors, and mortality, especially for stroke, compared to the general population. From 1994-2003 stroke mortality in ANAIs was at least 25% higher than for Whites in Alaska. Over the same period, stroke mortality for ANAIs under age 45 increased 400%, but declined in Whites. In addition, the decline in age-adjusted CVD mortality observed in recent decades within the general population does not extend to ANAIs. Controlling hypertension is a pillar of prevention for CVD and stroke.

Although ANAIs were formerly thought to have a very low prevalence of stroke and CVD, more reliable newer data indicate high levels of hypertension and associated mortality. A recent systematic review of 141 publications on hypertension in ANAI people documented a significant increase in recorded prevalence over the past 3 decades, as well as a significantly higher prevalence in ANAI adults than in reference populations, usually White. Aggregated data from the Behavioral Risk Factor Surveillance System (BRFSS) also show a higher prevalence of self-reported hypertension in ANAIs than in non-Hispanic Whites (27% vs. 22%). The National Health Interview Survey found a similar disparity of 35% vs 26% in ANAIs vs. Whites. As in non-Hispanic Whites, 61% of ANAIs with hypertension were taking anti-hypertensive medication. In a previous study, an investigator on the present proposal examined the health records of 524 ANAI elders, finding that 23% had undiagnosed hypertension, and 38% had diagnosed hypertension. Of those with diagnoses, 81% were taking medication, 37% had well-controlled blood pressure (BP), and lifestyle counseling was rare.

Ongoing management of high BP often requires healthcare providers to initiate or intensify therapy in response to uncontrolled high BP. A recent review concluded that the patient/provider relationship, patient/provider communication, and patient-centered decision making were essential to appropriate decisions on medication change. Another study using electronic health record (EHR) data on military veterans found that ~60% of patients with hypertension had poorly controlled systolic BP, yet less than half of clinicians made medication changes after a computer-generated notification.

Improving BP control requires the involvement not only of individuals but of healthcare systems and social environments. Communications must extend care to patients "where patients are" outside the clinic; facilitate BP self-management; and minimize barriers to care AN/AIs face in healthcare access. Across Alaska, 60% of residents are medically underserved, and in 75% of Alaskan communities, regardless of residents' race, comprehensive healthcare services are accessible only by air or water. Even in urban areas, health disparities among AN/AIs persist, and access to care is affected by factors such as lack of transportation.

CVD morbidity, mortality, and organ damage are more accurately predicted by home blood pressure monitoring (HBPM) than by in-office measurements. HBPM avoids over-treating sporadic high BP readings and "white coat" hypertension while facilitating control of both resistant and "masked" hypertension (high at home and normal in the clinic), which are associated with stroke. Compared to usual care or HBPM alone, HBPM combined with self-titration of medications or with physician, pharmacist, or nurse management leads to better use of medications and BP control. Research shows the value of using HBPM values to trigger modifications in anti-hypertensive regimens, and the addition of provider feedback, patient and provider education, and decision-making support to encourage treatment adjustments improves control even more. HBPM can support patient decision making, provide data to providers, facilitate patient/provider communication, and engage, educate, and empower patients. HBPM devices are widely accepted by patients, who prefer them to clinic-based measurements. HBPM interventions appear to be most effective in patients with less well-controlled BP at baseline. Therefore, tailored HBPM interventions have been developed for minorities, who may receive more benefit from HBPM than Whites.

Significance:

BP-ICAN is innovative in many ways. First, it will be the only rigorous, population-based study about BP control for prevention of CVD and stroke in ANs, and one of very few multilevel interventions in any minority population. Second, the Southcentral Foundation (SCF) service area includes rural, suburban, and urban locations. Third, the intervention design addresses therapeutic inertia, a well-recognized barrier to hypertension control that is often neglected in clinical trials, so the approach to improve self-efficacy and ownership should lead to more timely communication with providers and titration of medications.

The investigators will conduct a group-randomized trial for improving BP control among ANAI adults with diagnosed hypertension. Study group assignment will occur by randomizing all SCF primary care panels to the BP-ICAN or usual care control arms; adults with uncontrolled hypertension will be nested within groups defined by panel, which corresponds to one provider. For each panel, investigators will recruit up to 10 ANAI adults (expecting average of 8-9 per provider, for a total n = 324) who have had systolic BP ≥ 130 mmHg measured at one or more clinic visits in the past 18 months OR who have previously diagnosed hypertension and systolic BP ≥ 130 mmHg measured at the study screening or home screening visit. The study period for all participants will last 12 months.

Participants who are randomized to the BP-ICAN arm will receive education about BP control, CVD and stroke and the importance of hypertension management for prevention, other lifestyle changes that can prevent or reduce morbidity from hypertension, and educational materials about the importance of timely response to uncontrolled hypertension. BP-ICAN arm participants will also receive HBPM equipment (Omron device) and training in its use, interpretation of results, and assistance with communicating high BP values to healthcare providers. Lastly, participants will receive culturally tailored text messages to reinforce the educational material and motivate adherence to HBPM and provider communication strategies. Participants whose providers have been randomized to the control condition will continue to receive care as usual.

Patient-initiated communication about uncontrolled BP will serve as one component of the provider-level intervention. Participants will be trained to sync HBPM and smart phone to automatically upload BP measurements into a data repository using Omron's free wellness application. This will update the participant's data on Omron's Wellness Application website. Investigators plan to use a cloud-based technology platform to serve as a data repository and are working with tribal leadership, institutional privacy officers, compliance officers, and providers on how data will displayed and stored within the health care system. The goal is to make aggregate BP measure data available to providers in either a personal health record (PHR) and/or health information exchange (HIE) that allows for transmission of select measures into the electronic health and or population health record. Note that this protocol was developed based on extensive collaboration with SCF providers.

At the individual level, the primary outcome is within-person change in systolic BP. Secondary outcomes are diastolic BP, anti-hypertensive medication use and adherence, physical activity, weight, and tobacco use. Individual-level outcomes will be measured at baseline, 3 months, 6 months, and 1 year post-baseline. At the provider level, the primary outcome is change in prescribing behavior for medication and other relevant lifestyle changes. At the systems level, the primary outcome is change in systolic BP for all adults with hypertension whose providers are randomized to the BP-ICAN arm vs. the care as usual arm, regardless of whether the adults were directly enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least one visit to SCF providers or Community Health Aides within the previous year
2. Alaska Native or American Indian
3. At least 18 years old
4. Meet one of the following two conditions:

   I. Hypertension diagnosis and 1 systolic blood pressure (SBP) >= 140 mmHg in past 24 months in EHR, AND
   1. SBP >= 140 mmHg at research visit or from the mean of BP measures during the home screening period, OR
   2. SBP 130-139 mmHg at research visit or from the mean of BP measures during the home screening period plus at least one comorbid condition as stated in American Heart Association guidelines (cardiovascular disease, heart failure, stroke, atrial fibrillation, chronic kidney disease, kidney transplant, or diabetes) II. No hypertension diagnosis but 1 SBP >= 140 mmHg in past 18 months in EHR, AND

   <!-- -->

   1. SBP >=140mmHg at research visit or from the mean of BP measures during the home screening period, OR
   2. SBP 130-139 mmHg at research visit or from the mean of BP measures during the home screening period plus at least one comorbid condition as stated in AHA guidelines (cardiovascular disease, heart failure, stroke, atrial fibrillation, chronic kidney disease, kidney transplant, or diabetes)
5. Ability to provide informed consent
6. Willingness and ability to use a HBPM
7. Willingness to complete the necessary data collection procedures, including transmission of BP measurements and permission for study staff to access EHR and/or PHR data.

Exclusion criteria:

1. Does not meet inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Individual-level: within-person change in systolic blood pressure | 12 months
  Examine change in systolic blood pressure (mmHg) between participants in the intervention group compared to the control group.
Provider-level: frequency of antihypertensive medication adjustments | 3 months, 6 months, and 12 months
  Examine number of medication adjustments (new prescription or change in dose of antihypertensive medications) between participants in the intervention group compared to the control group.
System-level: change in systolic blood pressure for all patients with hypertension | 12 months
  Examine change in systolic blood pressure (mmHg) between all patients whose providers are in the intervention group (receiving automated alerts about high blood pressure and pharmacist support), compared to patients whose providers are in the control group (do not receive alerts and pharmacist support).

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Dillard, PhD, Principal Investigator — Southcentral Foundation
Locations (2):
- United States (2):
  - Anchorage Native Primary Care Center, Anchorage, Alaska
  - Benteh Nuutah Valley Native Primary Care Center, Wasilla, Alaska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris R, Nelson LA, Muller C, Buchwald D. Stroke in American Indians and Alaska Natives: A Systematic Review. Am J Public Health. 2015 Aug;105(8):e16-26. doi: 10.2105/AJPH.2015.302698. Epub 2015 Jun 11. PMID 26066955
- [Background] Hutchinson RN, Shin S. Systematic review of health disparities for cardiovascular diseases and associated factors among American Indian and Alaska Native populations. PLoS One. 2014 Jan 15;9(1):e80973. doi: 10.1371/journal.pone.0080973. eCollection 2014. PMID 24454685
- [Background] Jolly SE, Howard BV, Umans JG. Cardiovascular Disease Among Alaska Native Peoples. Curr Cardiovasc Risk Rep. 2013 Dec 1;7(6):10.1007/s12170-013-0362-5. doi: 10.1007/s12170-013-0362-5. PMID 24367710
- [Background] Howard BV, Devereux RB, Cole SA, Davidson M, Dyke B, Ebbesson SO, Epstein SE, Robinson DR, Jarvis B, Kaufman DJ, Laston S, MacCluer JW, Okin PM, Roman MJ, Romenesko T, Ruotolo G, Swenson M, Wenger CR, Williams-Blangero S, Zhu J, Saccheus C, Fabsitz RR, Robbins DC. A genetic and epidemiologic study of cardiovascular disease in Alaska natives (GOCADAN): design and methods. Int J Circumpolar Health. 2005 Jun;64(3):206-21. doi: 10.3402/ijch.v64i3.17985. PMID 16050315
- [Background] Horner RD, Day GM, Lanier AP, Provost EM, Hamel RD, Trimble BA. Stroke mortality among Alaska Native people. Am J Public Health. 2009 Nov;99(11):1996-2000. doi: 10.2105/AJPH.2008.148221. Epub 2009 Sep 17. PMID 19762671
- [Background] Trimble B, Morgenstern LB. Stroke in minorities. Neurol Clin. 2008 Nov;26(4):1177-90, xi. doi: 10.1016/j.ncl.2008.05.010. PMID 19026907
- [Background] Howard BV, Lee ET, Cowan LD, Devereux RB, Galloway JM, Go OT, Howard WJ, Rhoades ER, Robbins DC, Sievers ML, Welty TK. Rising tide of cardiovascular disease in American Indians. The Strong Heart Study. Circulation. 1999 May 11;99(18):2389-95. doi: 10.1161/01.cir.99.18.2389. PMID 10318659
- [Background] Foulds HJ, Warburton DE. The blood pressure and hypertension experience among North American Indigenous populations. J Hypertens. 2014 Apr;32(4):724-34. doi: 10.1097/HJH.0000000000000084. PMID 24609208
- [Background] Zhao G, Ford ES, Mokdad AH. Racial/ethnic variation in hypertension-related lifestyle behaviours among US women with self-reported hypertension. J Hum Hypertens. 2008 Sep;22(9):608-16. doi: 10.1038/jhh.2008.52. Epub 2008 May 22. PMID 18496555
- [Background] Barnes PM, Adams PF, Powell-Griner E. Health characteristics of the American Indian or Alaska Native adult population: United States, 2004-2008. Natl Health Stat Report. 2010 Mar 9;(20):1-22. PMID 20583451
- [Background] Rhoades DA, Buchwald D. Hypertension in older urban Native-American primary care patients. J Am Geriatr Soc. 2003 Jun;51(6):774-81. doi: 10.1046/j.1365-2389.2003.51261.x. PMID 12757563
- [Background] Rose AJ, Shimada SL, Rothendler JA, Reisman JI, Glassman PA, Berlowitz DR, Kressin NR. The accuracy of clinician perceptions of "usual" blood pressure control. J Gen Intern Med. 2008 Feb;23(2):180-3. doi: 10.1007/s11606-007-0464-1. Epub 2007 Nov 28. PMID 18043980
- [Background] Lebeau JP, Cadwallader JS, Aubin-Auger I, Mercier A, Pasquet T, Rusch E, Hendrickx K, Vermeire E. The concept and definition of therapeutic inertia in hypertension in primary care: a qualitative systematic review. BMC Fam Pract. 2014 Jul 2;15:130. doi: 10.1186/1471-2296-15-130. PMID 24989986
- [Background] Oakes JM. The (mis)estimation of neighborhood effects: causal inference for a practicable social epidemiology. Soc Sci Med. 2004 May;58(10):1929-52. doi: 10.1016/j.socscimed.2003.08.004. PMID 15020009
- [Background] Diez Roux AV. Complex systems thinking and current impasses in health disparities research. Am J Public Health. 2011 Sep;101(9):1627-34. doi: 10.2105/AJPH.2011.300149. Epub 2011 Jul 21. PMID 21778505
- [Background] Bobrie G, Chatellier G, Genes N, Clerson P, Vaur L, Vaisse B, Menard J, Mallion JM. Cardiovascular prognosis of "masked hypertension" detected by blood pressure self-measurement in elderly treated hypertensive patients. JAMA. 2004 Mar 17;291(11):1342-9. doi: 10.1001/jama.291.11.1342. PMID 15026401
- [Background] Niiranen TJ, Hanninen MR, Johansson J, Reunanen A, Jula AM. Home-measured blood pressure is a stronger predictor of cardiovascular risk than office blood pressure: the Finn-Home study. Hypertension. 2010 Jun;55(6):1346-51. doi: 10.1161/HYPERTENSIONAHA.109.149336. Epub 2010 Apr 12. PMID 20385970
- [Background] Stergiou GS, Christodoulakis GR, Nasothimiou EG, Giovas PP, Kalogeropoulos PG. Can validated wrist devices with position sensors replace arm devices for self-home blood pressure monitoring? A randomized crossover trial using ambulatory monitoring as reference. Am J Hypertens. 2008 Jul;21(7):753-8. doi: 10.1038/ajh.2008.176. Epub 2008 Apr 24. PMID 18443566
- [Background] Viera AJ, Lin FC, Tuttle LA, Olsson E, Stankevitz K, Girdler SS, Klein JL, Hinderliter AL. Reproducibility of masked hypertension among adults 30 years or older. Blood Press Monit. 2014 Aug;19(4):208-15. doi: 10.1097/MBP.0000000000000054. PMID 24842491
- [Background] Ohkubo T, Asayama K, Kikuya M, Metoki H, Obara T, Saito S, Hoshi H, Hashimoto J, Totsune K, Satoh H, Imai Y. Prediction of ischaemic and haemorrhagic stroke by self-measured blood pressure at home: the Ohasama study. Blood Press Monit. 2004 Dec;9(6):315-20. doi: 10.1097/00126097-200412000-00009. PMID 15564987
- [Background] Asayama K, Ohkubo T, Kikuya M, Metoki H, Hoshi H, Hashimoto J, Totsune K, Satoh H, Imai Y. Prediction of stroke by self-measurement of blood pressure at home versus casual screening blood pressure measurement in relation to the Joint National Committee 7 classification: the Ohasama study. Stroke. 2004 Oct;35(10):2356-61. doi: 10.1161/01.STR.0000141679.42349.9f. Epub 2004 Aug 26. PMID 15331792
- [Background] McManus RJ, Mant J, Bray EP, Holder R, Jones MI, Greenfield S, Kaambwa B, Banting M, Bryan S, Little P, Williams B, Hobbs FD. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010 Jul 17;376(9736):163-72. doi: 10.1016/S0140-6736(10)60964-6. Epub 2010 Jul 8. PMID 20619448
- [Background] Parati G, Omboni S, Albini F, Piantoni L, Giuliano A, Revera M, Illyes M, Mancia G; TeleBPCare Study Group. Home blood pressure telemonitoring improves hypertension control in general practice. The TeleBPCare study. J Hypertens. 2009 Jan;27(1):198-203. doi: 10.1097/hjh.0b013e3283163caf. PMID 19145785
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] Brennan T, Spettell C, Villagra V, Ofili E, McMahill-Walraven C, Lowy EJ, Daniels P, Quarshie A, Mayberry R. Disease management to promote blood pressure control among African Americans. Popul Health Manag. 2010 Apr;13(2):65-72. doi: 10.1089/pop.2009.0019. PMID 20415618
- [Background] Omboni S, Guarda A. Impact of home blood pressure telemonitoring and blood pressure control: a meta-analysis of randomized controlled studies. Am J Hypertens. 2011 Sep;24(9):989-98. doi: 10.1038/ajh.2011.100. Epub 2011 Jun 9. PMID 21654858
- [Background] Roumie CL, Elasy TA, Greevy R, Griffin MR, Liu X, Stone WJ, Wallston KA, Dittus RS, Alvarez V, Cobb J, Speroff T. Improving blood pressure control through provider education, provider alerts, and patient education: a cluster randomized trial. Ann Intern Med. 2006 Aug 1;145(3):165-75. doi: 10.7326/0003-4819-145-3-200608010-00004. PMID 16880458
- [Background] Carter BL, Ardery G, Dawson JD, James PA, Bergus GR, Doucette WR, Chrischilles EA, Franciscus CL, Xu Y. Physician and pharmacist collaboration to improve blood pressure control. Arch Intern Med. 2009 Nov 23;169(21):1996-2002. doi: 10.1001/archinternmed.2009.358. PMID 19933962
- [Background] Carter BL, Rogers M, Daly J, Zheng S, James PA. The potency of team-based care interventions for hypertension: a meta-analysis. Arch Intern Med. 2009 Oct 26;169(19):1748-55. doi: 10.1001/archinternmed.2009.316. PMID 19858431
- [Background] Hunt JS, Siemienczuk J, Pape G, Rozenfeld Y, MacKay J, LeBlanc BH, Touchette D. A randomized controlled trial of team-based care: impact of physician-pharmacist collaboration on uncontrolled hypertension. J Gen Intern Med. 2008 Dec;23(12):1966-72. doi: 10.1007/s11606-008-0791-x. Epub 2008 Sep 25. PMID 18815843
- [Background] Svetkey LP, Pollak KI, Yancy WS Jr, Dolor RJ, Batch BC, Samsa G, Matchar DB, Lin PH. Hypertension improvement project: randomized trial of quality improvement for physicians and lifestyle modification for patients. Hypertension. 2009 Dec;54(6):1226-33. doi: 10.1161/HYPERTENSIONAHA.109.134874. PMID 19920081
- [Background] Nasothimiou EG, Karpettas N, Dafni MG, Stergiou GS. Patients' preference for ambulatory versus home blood pressure monitoring. J Hum Hypertens. 2014 Apr;28(4):224-9. doi: 10.1038/jhh.2013.104. Epub 2013 Oct 24. PMID 24152822
- [Background] Bosworth HB, Powers BJ, Olsen MK, McCant F, Grubber J, Smith V, Gentry PW, Rose C, Van Houtven C, Wang V, Goldstein MK, Oddone EZ. Home blood pressure management and improved blood pressure control: results from a randomized controlled trial. Arch Intern Med. 2011 Jul 11;171(13):1173-80. doi: 10.1001/archinternmed.2011.276. PMID 21747013
- [Background] Kim MT, Han HR, Hedlin H, Kim J, Song HJ, Kim KB, Hill MN. Teletransmitted monitoring of blood pressure and bilingual nurse counseling-sustained improvements in blood pressure control during 12 months in hypertensive Korean Americans. J Clin Hypertens (Greenwich). 2011 Aug;13(8):605-12. doi: 10.1111/j.1751-7176.2011.00479.x. Epub 2011 Jun 27. PMID 21806771
- [Background] Odedosu T, Schoenthaler A, Vieira DL, Agyemang C, Ogedegbe G. Overcoming barriers to hypertension control in African Americans. Cleve Clin J Med. 2012 Jan;79(1):46-56. doi: 10.3949/ccjm.79a.11068. PMID 22219234
- [Background] Artinian NT, Flack JM, Nordstrom CK, Hockman EM, Washington OG, Jen KL, Fathy M. Effects of nurse-managed telemonitoring on blood pressure at 12-month follow-up among urban African Americans. Nurs Res. 2007 Sep-Oct;56(5):312-22. doi: 10.1097/01.NNR.0000289501.45284.6e. PMID 17846552
- [Background] Eby D. Integrated primary care. Int J Circumpolar Health. 1998;57 Suppl 1:665-7. PMID 10093362
- [Background] Mala TA, Gottlieb KL. Designing a home health care system for Alaska Natives in Anchorage. Int J Circumpolar Health. 1998;57 Suppl 1:675-8. PMID 10093365
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555

DOCUMENTS (1):
  • Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03872856/ICF_001.pdf